CLINICAL TRIAL: NCT04514237
Title: A Phase 1 Study to Determine the Relative Bioavailability of BOS172767 Enantiomer E1 and E2 and the Single and Repeat Dose Pharmacokinetics, Safety and Tolerability of BOS172767 Selected Enantiomer in Healthy Subjects
Brief Title: Study to Determine the Relative Bioavailability, Single and Repeat Dose Pharmacokinetics, Safety and Tolerability of BOS172767 Enantiomers in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: BOS172767-02; 2019-002289-11 (EudraCT Number); QSC201870 (Other: Quotient Sciences)
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Healthy Participants
Keywords: BOS172767; enantiomer E1 and E2; relative bioavailability; pharmacokinetics; dose linearity; healthy participants

STUDY DESIGN:
Intervention Model Description: Part 1 was a two-way crossover design, followed by two sequential ascending dose periods. Part 2 was designed to be a multiple ascending dose design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: Regimens AB(CD) (Experimental): Participants received 50 milligrams (mg) BOS172767 E1 tablets or matching placebo (Regimen A) in the fasted state in Period 1, followed by 50 mg BOS172767 E2 tablets or matching placebo (Regimen B) in the fasted state in Period 2. In Period 3 and 4, participants received BOS172767-Ex (selected enantiomer from Part 1 [E1 or E2]) tablets or matching placebo (Regimens C and D, respectively) from Regimen A or B in the fasted state. The Period 3 and 4 dose was selected after review of data from Periods 1 and 2. In each Period, dosing occurred on Day 1, and there was a washout period of at least 10 days or 5 half-lives of the parent (whichever is greater) between each dose of investigational medicinal product.
  Interventions: Drug: BOS172767 enantiomer E1 or E2; Drug: Placebo
- Part 1: Regimens BA(CD) (Experimental): Participants received 50 milligrams (mg) BOS172767 E2 tablets or matching placebo (Regimen B) in the fasted state in Period 1, followed by 50 mg BOS172767 E1 tablets or matching placebo (Regimen A) in the fasted state in Period 2. In Period 3 and 4, participants received BOS172767-Ex (selected enantiomer from Part 1 [E1 or E2]) tablets or matching placebo (Regimens C and D, respectively) from Regimen A or B in the fasted state. The Period 3 and 4 dose was selected after review of data from Periods 1 and 2. In each Period, dosing occurred on Day 1, and there was a washout period of at least 10 days or 5 half-lives of the parent (whichever is greater) between each dose of investigational medicinal product.
  Interventions: Drug: BOS172767 enantiomer E1 or E2; Drug: Placebo

INTERVENTIONS:
Drug: BOS172767 enantiomer E1 or E2 — Oral tablets
Drug: Placebo — Oral tablets

SUMMARY:
Part 1 of the study evaluates the safety and tolerability as well as pharmacokinetic properties of a single oral dose of BOS172767 enantiomer E1 and BOS172767 enantiomer E2 following administration to healthy participants. Part 2 of the study was to be conducted to assess the safety and tolerability as well as pharmacokinetic properties of one selected enantiomer (BOS172767-Ex) following multiple ascending doses over 14 days of dosing in healthy participants.

DETAILED DESCRIPTION:
The study design of Part 1 was a double-blind, placebo-controlled, randomized, single-dose, two-way crossover, followed by two sequential ascending dose periods in 12 healthy participants.

Part 2 was designed to be a double-blind, placebo-controlled, randomized multiple ascending dose (MAD) study in 36 healthy participants (12 per study cohort).

Part 2 was to progress following completion of Part 1, but was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy females of non-childbearing potential
* Age 18 to 50 years at the time of signing informed consent
* Body mass index (BMI) of 18.0 to 32.0 kilograms per meters squared (kg/m^2) as measured at screening
* Must have been willing and able to communicate and participate in the whole study
* Must have provided written informed consent
* Must have agreed to adhere to the contraception requirements for this study

Exclusion Criteria:

* Participants who received any investigational medicinal product (IMP) in a clinical research study within the 90 days prior to Day 1
* Participants who were study site employees, or immediate family members of a study site or sponsor employee
* Participants who had previously been enrolled and dosed in this study. Participants who had taken part in Part 1 were not permitted to take part in Part 2. Participants who had taken part in study QCL118174/BOS172767-01 (NCT03464058) were allowed to participate in this study.
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = 1/2 pint beer, or a 25 milliliter [mL] shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who had smoked within the last 6 months. A confirmed breath carbon monoxide reading of greater than 20 parts per million (ppm) at screening or admission.
* Current users of e-cigarettes and nicotine replacement products and those who had used these products within the last 6 months
* Females of childbearing potential including those who were pregnant or lactating (all female participants must have had a negative serum pregnancy test at screening and had a negative urine pregnancy test at all other time points). A woman was considered of childbearing potential unless she was permanently sterile (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) or was postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration ≥40 International Units per Liter [IU/L])
* Participants who did not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Clinically significant abnormal clinical chemistry, haematology, or urinalysis as judged by the investigator. Participants with Gilbert's Syndrome were not allowed.
* Participants with alanine aminotransferase (ALT) > 1.5 x upper limit of normal (ULN) at screening (Part 1 and Part 2) or Day -1 (Part 2 only)
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <70 milliliters per minute (mL/min) using the Cockcroft-Gault equation
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory, or gastrointestinal disease (including gall stones and/or cholecystectomy), or neurological or psychiatric disorder, as judged by the investigator
* Serious adverse reaction or serious hypersensitivity to any drug or the IMP excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever was allowed unless it was active.
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Participants who were taking, or had taken, any prescribed or over-the-counter drug (other than 4 grams of paracetamol per day and/or hormone replacement therapy [HRT]) or herbal remedies in the 14 days before IMP administration. Exceptions may have applied on a case by case basis, if considered not to have interfered with the objectives of the study, as determined by the principal investigator.
* Participants who had any ongoing fungal infections (stable toe nail onchomycosis was allowed)
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Part 1: Relative bioavailability of E1 versus E2 (Frel; exposure) of a single oral dose of BOS172767 enantiomer 1 (E1) and enantiomer 2 (E2) following administration to healthy participants based on Cmax, AUC(0-last), and AUC (0-inf) | 24 hours post-dose for each of the four 6-day Periods
  Cmax is defined as the maximum observed concentration. AUC(0-last) is defined as the area under the curve from 0 time to the last measurable concentration. AUC (0-inf) is defined as the area under the curve from 0 time extrapolated to infinity.
Part 1: Number of participants with any treatment-emergent adverse event | up to Day 6 of each Period; up to a 10-day Follow-up Period after last dose (up to Study Day 59)
Part 1: Number of participants with abnormal, clinically significant physical examination findings | up to Day 6 of each Period; up to a 10-day Follow-up Period after last dose (up to Study Day 59)
Part 1: Number of participants with abnormal, clinically significant safety laboratory test findings | up to Day 6 of each Period; up to a 10-day Follow-up Period after last dose (up to Study Day 59)
Part 1: Number of participants with abnormal, clinically significant vital sign values | up to Day 6 of each Period; up to a 10-day Follow-up Period after last dose (up to Study Day 59)
Part 1: Number of participants with abnormal, clinically significant electrocardiogram findings | up to Day 6 of each Period; up to a 10-day Follow-up Period after last dose (up to Study Day 59)
Part 1: Plasma concentration of BOS172767 enantiomers 1 and 2 | 24 hours post-dose for each of the four 6-day Periods
Part 1: Slope estimates (β) from the power model analysis on Cmax, AUC(0-last), and AUC(0-inf), as a measure of dose proportionality | 24 hours post-dose for each of the four 6-day Periods
Part 2: Plasma concentration of BOS172767-Ex (enantiomer E1 or E2) | 24 hours post-dose
Part 2: Number of participants with any treatment-emergent adverse event | up to Day 24 of Part 2 (up to approximately 18 study weeks)
Part 2: Number of participants with abnormal, clinically significant physical examination findings | up to Day 24 of Part 2 (up to approximately 18 study weeks)
Part 2: Number of participants with abnormal, clinically significant safety laboratory test findings | up to Day 24 of Part 2 (up to approximately 18 study weeks)
Part 2: Number of participants with abnormal, clinically significant vital sign values | up to Day 24 of Part 2 (up to approximately 18 study weeks)
Part 2: Number of participants with abnormal, clinically significant electrocardiogram findings | up to Day 24 of Part 2 (up to approximately 18 study weeks)
Part 2: Slope estimates (β) from the power model analysis on Cmax, AUC(0-last), and AUC(0-inf), as a measure of dose proportionality | 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No